

Version number and date: 06/11/2023 (2)

[IRAS ID: 330859]

## **CONSENT FORM**

| Title | ٥f | study | /· F | reP | -ACe |
|-------|----|-------|---------|-----|------|
| 11110 | vı | Stuui | / . I | 101 | -706 |

Name of Researcher: Dr Sarah Raut, Prof Lee Ingle, Prof Gerard Danjoux, Dr Simon Davies, Dr David

| Yates | | |
|---|---|---|
| | | Please initial box |
| 1.I confirm that I have read the information sheet dated 06/11/2023 version 4 for the<br>above study. I have had the opportunity to consider the information, ask questions and have<br>had any questions answered satisfactorily. | | |
| without giving any re | eason, without my medical c | I that I am free to withdraw at any time care or legal rights being affected. I the point of withdrawal will be retained. |
| the study, may be a from the NHS Trust | ccessed by individuals from | aking part in this research. I give permission for |
| | research data, which will be<br>I publicly disseminated. | anonymised (not linked to me), will be retained by |
| 5.I understand that my of the future. (optional | _ | be shared with others to support other research in |
| • • | personal data will be kept se<br>ally be available to the immed | ecurely in accordance with data protection diate research team |
| 7. I give permission for the research question | he collection and use of my on in this study. | data to answer |
| 8.I agree to take part in | the above study. | |
| Name of Participant | <br>Date | Signature |
| Name of Person taking consent | Date | Signature |



9.I agree for my data to be shared with other researchers to support future research.

Name of Participant

Date

Signature

Name of Person

Date

Signature

taking consent